CLINICAL TRIAL: NCT03346941
Title: Side Effects After Direct-acting Antiviral Treatment in Patients With Chronic Hepatitis C. The EFINO-C Study.
Brief Title: Side Effects After Direct-acting Antiviral Treatment
Acronym: EFINO-C
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_004
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: DAA treatment — Direct-acting antiviral-based treatment

SUMMARY:
The objective of this study was to assess the incidence of side effects after direct-acting antiviral therapy in patients with chronic hepatitis C virus infection.

DETAILED DESCRIPTION:
Direct-acting antiviral (DAA)-based treatments are today very effective The objective of this study was to assess the incidence of side effects after DAA therapy in patients with chronic hepatitis C virus infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Hepatitis C virus infection
* Treatment by direct-acting antiviral combination

Exclusion Criteria:

* HIV coinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with direct-acting antiviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of side effects | Within treatment duration, i.e. 8, 12 or 24 weeks after treatment initiation
  Incidence of side effects occurring during treatment duration. Treatment duration may be of 8 weeks, 12 weeks or 24 weeks depending on treatment combination.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No